CLINICAL TRIAL: NCT04404036
Title: Treatment of Eustachian Tube Dysfunction (ETD) and Facial Pain With Combined Acoustic Vibration and Oscillating Expiratory Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Shaun A. Nguyen, MD, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO#00097842
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Eustachian Tube Dysfunction; Facial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SinuSonic Device (Experimental): Aim 1: SinuSonic device used once a day over a 2 day period.
  Aim 2: SinuSonic device used twice daily for 3 minutes in the home setting for 6 weeks.
  Aim 3: SinuSonic device used twice daily for 3 minutes in the home setting for 4 weeks.
  Interventions: Device: SinuSonic Device

INTERVENTIONS:
Device: SinuSonic Device — A medical device that utilizes sound and pressure combined with normal breathing to relieve nasal congestion.

SUMMARY:
This study aims to test the safety, efficacy and potential mechanism of action of the SinuSonic device on adults with eustachian tube dysfunction (ETD) or facial pain/pressure. SinuSonic is a medical device that utilizes sound and pressure combined with normal breathing. The study will have 3 aims. Aim 1 will examine healthy controls with no signs of upper respiratory infection, inflammation, or ETD to determine if exhaled nasal Nitric Oxide is increased. Nitric Oxide is a compound in the body that acts as a blood vessel relaxant. Acoustic energy (humming) has been shown to increase nasal Nitric Oxide dramatically, thus equalization of gas pressures between the middle ear, the paranasal sinuses and the nasal cavity may very well explain any efficacy noted. Aim 2 will be performed to examine therapeutic efficacy for ETD. Aim 3 will be performed to examine therapeutic efficacy for sinus pain/pressure.

ELIGIBILITY:
AIM 1

Inclusion Criteria:

* Adults 18 years or older with no symptoms of URI, ETD or other ENT conditions

Exclusion Criteria:

* Sinonasal or ear surgery within last 3 months (including balloon ET dilation)
* Any ENT condition that may impact upper airway to include sinusitis, otitis, or allergies
* Upper respiratory illness within last 2 weeks
* Topical decongestant use in last week
* Current nasal crusting or ulceration on rhinoscopy
* History of severe nose bleeding within last 3 months
* Known pregnancy
* Allergic sensitivity to silicone or any other component of device
* Inability to read and understand English
* Inability to perform treatment due to underlying medical condition

AIM 2

Inclusion:

* Adults 18 years or older with diagnosis of ETD by an otolaryngologist
* ≥6 months of symptoms duration
* ≥3 ETD symptoms (ear pressure, feeling that ears are clogged, cracking/popping of ears, muffled hearing, tinnitus)
* ETDQ-7 score ≥ 3
* Audiogram within the last year

Exclusion:

* Sinonasal or ear surgery within last 3 months (including balloon ET dilation)
* Indwelling ear tubes
* Tympanic membrane perforation
* Hx of cholesteatoma, mastoidectomy, tympanoplasty, or ossicular chain reconstruction
* Patulous ET
* Hx of Meniere's disease
* Moderate or severe nasal valve collapse
* Grade 3-4 polyps
* Upper respiratory illness within last 2 weeks
* Topical decongestant use in last week
* Current nasal crusting or ulceration on rhinoscopy
* History of severe nose bleeding within last 3 months
* Known pregnancy
* Allergic sensitivity to silicone or any other component of device
* Inability to read and understand English
* Inability to perform treatment due to underlying medical condition

AIM 3

Inclusion:

* Adults 18 years or older who complain of facial pain or pressure
* ≥3 months of symptoms duration (can be intermittent)
* Pain/pressure VAS score ≥ 5

Exclusion:

* Sinonasal surgery within the last 3 months
* Grade 3-4 polyps
* Upper respiratory illness within last 2 weeks
* Topical decongestant use in last week
* Current nasal crusting or ulceration on rhinoscopy
* History of severe nose bleeding within last 3 months
* Known pregnancy
* Allergic sensitivity to silicone or any other component of device
* Inability to read and understand English
* Inability to perform treatment due to underlying medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Symptoms severity according to an ETD Visual Analogue Scale | 6 Weeks
  Symptoms severity will be assessed on Visual Analogue Scale (on the scale of 1-10). Visual Analogue Scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Symptoms severity according to a Pain/pressure Visual Analogue Scale | 2 to 4 Weeks
  Symptoms severity will be assessed on Visual Analogue Scale (on the scale of 1-10). Visual Analogue Scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.

SECONDARY OUTCOMES:
McGill Pain Questionnaire - Short Form | 2 to 4 Weeks
  The MPQ-SF is a well-validated pain measure that permits separation of the sensory and affective components of pain, which are averaged to compute a total score. The scale ranges from 0-10 (0=no pain, 10=the most pain).
Worst Pain Using the Modified Brief Pain Inventory - Short Form (m-BPI-sf) | 2 to 4 Weeks
  Modified Brief Pain Inventory - Short Form (m-BPI-sf): participant rated 11-point Likert rating scale ranged from 0 (no pain) to 10 (worst pain imaginable).
Mean Change in Overall ETDQ-7 Score | 6 Weeks
  Mean change from baseline to 6 weeks in the overall ETDQ-7 score. The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that the participant's ears are clogged or underwater, ear symptoms when the participants have a cold or sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that the participant's hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinus Center - Medical Univesity of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Not Applicable. The investigators plan to publish this study.